CLINICAL TRIAL: NCT01282710
Title: Comparison of SureCALL® EMG Labor Monitor® and Tocodynamometer to Intrauterine Pressure Catheter Measurement in Pregnant Women
Brief Title: Comparison of SureCALL® EMG Labor Monitor® and Tocodynamometer to Intrauterine Pressure Catheter Measurement (IUPC) Measurement in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Reproductive Research Technologies, LP (Industry)
Responsible Party: Jack McCrary, Managing Director, Reproductive Research Technologies, LP
Other Study IDs: RRT-09-01
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-02

CONDITIONS: Pregnancy - Labor Monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Pregnant, In Labor

SUMMARY:
This measurement study was designed to evaluate the performance of SureCALL® EMG Labor Monitor® (SureCALL®) to the predicate Tocodynamometer device (TOCO) using the performance of an Intrauterine Pressure Catheter device (IUPC) as the "gold standard".

DETAILED DESCRIPTION:
The SureCALL® EMG Labor Monitor® (SureCALL®) is a transabdominal electromyography monitor intended to measure intrapartum uterine activity. It is intended for use on term pregnant women who are in labor, with singleton pregnancies, using surface electrodes on the maternal abdomen. The device is intended for use by healthcare professionals in a clinical setting.

This measurement study was designed to evaluate the performance of SureCALL® to the predicate Tocodynamometer device (TOCO) using the performance of an Intrauterine Pressure Catheter device (IUPC) as the "gold standard".

This study involved 20 women at term, in labor, at three clinical sites. Each study subject was instrumented with three technologies for measuring uterine activity:

1. a tocodynamometer attached to the maternal abdomen
2. a set of abdominal surface electrodes for uterine electromyography, and
3. an intrauterine pressure catheter.

Using IUPC as the "gold standard", this study methodology allowed a three way comparison for evaluating how well the SureCALL® system performed compared to the TOCO technology.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy
* Indicated for IUPC
* Gestational ages from 37 to 41 weeks
* Informed consent required

Exclusion Criteria:

* Multifetal Pregnancy
* Not Indicated for IUPC
* Gestation ages below 37 or above 41 weeks
* Informed consent not given

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women in labor with uncomplicated singleton pregnancies and IUPC indicated with membranes ruptured and sufficient cervical dilation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Waterhouse, MD, Principal Investigator — Reproductive Research Technologies, LP
Locations (3):
- United States (3):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregnant, In Labor: Monitored simultaneously by SureCALL®, TOCO, and IUPC
Period: Overall Study
Arm/Group | Pregnant, In Labor
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pregnant, In Labor
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.85 (4.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Comparison of SureCALL® and TOCO Detection of Contraction Events, as Compared to the IUPC
Description: Contraction timing as measured by the SureCALL® and contraction timing as measured by the TOCO, both compared to the contraction timing as measured by the IUPC gold standard. The contraction timing values of SureCALL® and TOCO were then compared.
Time Frame: 9 - 42 Minutes
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Pregnant, In Labor
Number analyzed (Participants) | 20
Seconds
  SureCALL® and IUPC Peak Time Difference | -0.73 (9.22)
  TOCO and IUPC Peak Time Difference | -1.74 (8.25)
Statistical Analysis 1: Comparison: Pregnant, In Labor; Agreement between SureCALL® and IUPC Contraction Peak Events Null hypothesis: the mean peak difference between TOCO and IUPC is equal to 0. Alternative hypothesis: the mean peak difference is not equal to 0; Test type: Superiority or Other; p = .04627, Mixed Models Analysis
Statistical Analysis 2: Comparison: Pregnant, In Labor; Agreement between TOCO and IUPC Contraction Peak Events Null hypothesis: the mean peak difference between TOCO and IUPC is equal to 0. Alternative hypothesis: the mean peak difference is not equal to 0; Test type: Superiority or Other; p = 0.1676, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Pregnant, In Labor
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs may publish or present results of the study after the expiration of 12 months from completion. Publications or presentations are subject to the protection of confidential information or patentable information.